CLINICAL TRIAL: NCT03289117
Title: Evaluation of a Novel Medical Device to Facilitate Gel Instillation During Change of Long-term Indwelling Urinary Catheters - a Randomized Controlled Study
Brief Title: Evaluation of a Novel Medical Device to Facilitate Gel Instillation During Change of Long-term Urinary Catheters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other); Vinnova (Other Government); Innovation Skåne AB/ Sweden (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2016 02 01 ver 1_1
Record Dates: First submitted 2017-09-18; First posted 2017-09-20 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Urinary Catheters; Retention, Urinary; Incontinence, Urinary; Anesthesia, Local
Keywords: Urinary catheterization; Gel installation; Novel medical device; Indwelling urinary catheter; Long-term urinary catheter; Male patients
MeSH Terms: conditions — Urinary Retention; Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: Arm 1: Experimental: Novel device: Assigned Interventions: Catheter change with novel device. Each subject will undergo catheter change with novel gel instillation device.
  Arm 2: Comparator: Standard procedure: Assigned Interventions: Catheter change with standard procedure. Each subject will undergo catheter change with standard procedure.
Who Masked: Outcomes Assessor
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Novel gel installation device procedure (Experimental): Catheter change with novel device.
  Each subject will undergo catheter change with novel gel instillation device procedure
  Interventions: Device: Novel gel installation device procedure
- Standard procedure (Active Comparator): Catheter change with standard procedure.
  Each subject will undergo catheter change with standard procedure
  Interventions: Device: Standard procedure

INTERVENTIONS:
Device: Novel gel installation device procedure — Catheter change with novel device Each subject will undergo catheter change with novel gel instillation device
  Arms: Novel gel installation device procedure
Device: Standard procedure — Catheter change with standard procedure Each subject will undergo catheter change with standard procedure
  Arms: Standard procedure

SUMMARY:
A randomized, open label, controlled, parallel group study to investigate difference between regional standard procedure and a novel modified procedure (using an additional novel device to facilitate gel installation) for changing long-term indwelling urinary catheters.

DETAILED DESCRIPTION:
This is a randomized, open label, controlled, parallel group study, which comprises one visit that includes: assessment for eligibility, randomization to one of two treatment alternatives, followed by the actual intervention and evaluation of outcomes.

The interventions are either change of catheter according to the regional standard procedure (the comparator group) or change of catheter with the additional use of the novel device to facilitate gel instillation and a slightly modified procedure (the experimental group).

ELIGIBILITY:
Inclusion Criteria:

* The patient has an indwelling catheter and a primary diagnosis that justify continued catheter use
* The patient provides informed consent prior to any study specific procedures
* The patient is considered to benefit from participation in the clinical study

Exclusion Criteria:

* The patient do not consent to participate in the study
* Trauma to urethra or bladder
* Infection to urethra or bladder
* Other diagnosis that contraindicates participation in the clinical study as judged by the responsible physician

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-04-17 (Actual); Primary Completion 2017-05-26 (Actual); Study Completion 2017-05-26 (Actual)

PRIMARY OUTCOMES:
Treatment duration (min) | During procedure
  Treatment duration for procedure

SECONDARY OUTCOMES:
Patient's perceived pain (NRS scale) | During intervention
  Patient's perceived pain estimated by patient using a numerical rating scale (NRS-scale)
Number of gel syringes used | During intervention
  Number of pre-filled gel syringes used during the procedure

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | During intervention
  Incidence of Treatment-Emergent Adverse Events found during procedure

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Malmqvist, PhD, Principal Investigator — Clinical Studies Sweden - Forum South
Locations (1):
- Skåne University Hospital - Urology clinic - Homecare unit, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No